CLINICAL TRIAL: NCT04123379
Title: Tisch Cancer Institute - BMS Study # CA027-005: Neoadjuvant Nivolumab + BMS-813160 (CCR2/5-inhibitor) or BMS-986253 (anti-IL-8) for NSCLC or HCC
Brief Title: Neoadjuvant Nivolumab with CCR2/5-inhibitor or Anti-IL-8) for Non-small Cell Lung Cancer (NSCLC) or Hepatocellular Carcinoma (HCC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Thomas Marron, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-1754
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer; Hepatocellular Carcinoma
Keywords: Nivolumab; CCR2/5-inhibitor; anti-IL-8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular | interventions — Nivolumab; BMS-813160; HuMax-IL8

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A (Experimental): NSCLC: Nivolumab + BMS-813160
  Interventions: Drug: Nivolumab; Drug: BMS-813160
- Cohort B (Experimental): NSCLC: Nivolumab + BMS-986253
  Interventions: Drug: Nivolumab; Drug: BMS-986253
- Cohort C (Experimental): HCC: Nivolumab
  Interventions: Drug: Nivolumab
- Cohort D (Experimental): HCC: Nivolumab + BMS-813160
  Interventions: Drug: Nivolumab; Drug: BMS-813160
- Cohort E (Experimental): HCC: Nivolumab + BMS-986253
  Interventions: Drug: Nivolumab; Drug: BMS-986253

INTERVENTIONS:
Drug: Nivolumab — q4w, dosed twice before surgery and three times following recovery from surgery by injection
Drug: BMS-813160 — 300mg oral twice a day for 28 days
  Other Names: CCR2/5-inhibitor
  Arms: Cohort A; Cohort D
Drug: BMS-986253 — 2400mg once by injection
  Other Names: anti-IL-8
  Arms: Cohort B; Cohort E

SUMMARY:
The purpose of this research study is to study the effect of giving nivolumab with CCR2/5-inhibitor or anti-IL-8 before surgery, and after surgery, with the goal of determining if this medicine results in:

1. A significant immune response against their tumor (which the study team will see in the tumor that is taken out at the time of surgery)
2. Improvement in long term survival rates

DETAILED DESCRIPTION:
Objectives:

Cohorts A,B (NSCLC):

Primary Objective: Major Pathologic Response (MPR) Secondary Objectives: Time to surgery, tolerability and safety, radiographic response

Cohorts C,D,E (HCC):

Primary Objective: Significant tumor necrosis (STN) Secondary Objectives: Time to surgery, tolerability and safety, radiographic response

Diagnosis and Main Inclusion Criteria:

Patients must have disease deemed resectable before enrollment.

Study Product:

Nivolumab 480mg (q4w, dosed twice before surgery and three times following recovery from surgery) BMS-813160 (CCR2/5-inhibitor) 300mg oral twice a day for 28 days BMS-986253 (anti-IL-8) 2400mg once

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSCLC or HCC
* Willing to provide blood samples
* Willing to undergo leukapheresis at Mount Sinai Hospital or New York Blood Bank
* Willing to have excisional or core needle biopsies
* At least 18 years of age
* ECOG 0-1
* Surgical candidate for resection of their tumor
* Agree to use adequate contraception
* Adequate organ and marrow function

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 months for a different primary tumor or patients who have received locoregional therapy for the target lesion
* Patients receiving any other investigational agents
* Patients with metastatic disease for whom the intent of surgery would not be curative
* Uncontrolled intercurrent illness
* Pregnant or nursing
* Has a diagnosis of primary immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days
* Has active autoimmune disease that has required systemic treatment in the past year
* Has a known additional malignancy that is progressing and/or requires active treatment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not the in the best interest of the patient to participate
* HIV positive with detectable viral load or anyone not on stable anti-viral regimen
* Has known active Hepatitis B
* History of allogeneic hematopoietic cell transplantation or solid organ transplantation
* Documented allergic or hypersensitivity response to any protein therapeutics
* Patients may not have prolonged QRS or QTc

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) | 2 Years
  MPR is defined as <10% viable tumor within resection, at time of surgery.
Significant Tumor Necrosis (STN) | 2 Years
  STN is defined as necrosis of >70% of tumor base on pathologic analysis of gross tumor resection at time of surgery.

SECONDARY OUTCOMES:
Time to Surgery | 2 Years
  Measured as the time in days that elapses between the first dose of neoadjuvant therapy and surgical resection.
Percent of individuals who experience adverse events | 2 Years
  Safety and Tolerability defined by the percent of individuals who experience adverse events at any point during the neoadjuvant period, or within 30 days following the final dose of nivolumab received.
Percent of individuals who experience radiographic response | 2 Years
  As per RECIST v1.1 as determined by pre-surgical imaging, following receipt of the neoadjuvant therapy. For NSCLC this will be based on CT imaging, while for HCC this imaging will be based on MRI radiographic post-contract subtraction.
Progression-free survival (PFS) | 2 Years
  Defined as the time, in days, between treatment initiation and when the patient is found to have recurrent and/or metastatic disease on imaging, or death for any reason.
Overall Survival (OS) | 2 Years
  Defined as the time, in days, between treatment initiation and when the patient dies from any cause regardless of etiology.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marron, MD PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States